CLINICAL TRIAL: NCT06107010
Title: Effects of Atalante Exoskeleton on Gait Recovery in Non- or Poorly Ambulatory Patients With Hemiparesis in the Acute/Subacute Phase (Month 1 to 4)
Acronym: EarlyExo
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EarlyExo
Record Dates: First submitted 2023-10-24; First posted 2023-10-30 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Stroke, Acute; Stroke, Ischemic; Stroke, Subacute; Stroke Hemorrhagic; Cerebrovascular Disorders; Cerebrovascular Accident; Hemiparesis; Hemiparesis;Poststroke/CVA; Hemiparesis/Hemiplegia (One Sided Weakness/Paralysis)
Keywords: Robotics; Rehabilitation; Powered Exoskeleton; Walking recovery; Stroke; Acute stroke; Subacute stroke; Functional Ambulation Category; Randomized controlled study
MeSH Terms: conditions — Stroke; Ischemic Stroke; Hemorrhagic Stroke; Cerebrovascular Disorders; Paresis; Hemiplegia

STUDY DESIGN:
Intervention Model Description: Single blind
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exo group (Experimental): During the 6-week intervention period, the Exo group will complete 3 sessions per week (i.e., 18 one-hour sessions) with the Atalante device and 2 sessions per week (i.e., 12 one-hour sessions) of conventional therapy.
  During sessions with the exoskeleton, the patient will perform ambulatory exercises with the device, with a gradual increase of intensity through the sessions.
  Conventional therapy corresponds to physiotherapy as part of post stroke standard of care of the center (tasks such as lower and upper limb practice, walking in parallel bars, etc., but this list is not exhaustive and depends on the practice of the therapists/centers).
  Interventions: Device: Use of the Atalante exoskeleton
- Control group (No Intervention): During the 6-week intervention period, the Control group will complete 5 sessions per week of conventional therapy (i.e., 30 one-hour sessions).

INTERVENTIONS:
Device: Use of the Atalante exoskeleton — Six weeks of exoskeleton sessions replacing conventional therapy sessions three times a week
  Arms: Exo group

SUMMARY:
The present clinical investigation - EarlyExo, is an interventional, international, multicentric, prospective, single-blinded randomized controlled trial.

This clinical investigation is designed to test the hypothesis that early and intense introduction of walking sessions assisted by the Atalante exoskeleton, in a sample of hemiparetic patients with still non or poor ambulatory capacities (FAC 0 or 1) between one- and four-months post stroke, would result in a better recovery of functional walking compared to a control group only receiving conventional therapy. Improved recovery will be measured through the proportion of patients reaching a FAC score of 4 or higher at the end of the intervention period. The tested hypothesis is that this proportion will be higher in the Exo group.

The duration of the intervention period in both groups is 6 weeks.

* For the Exo group: 3 sessions per week (i.e., 18 one-hour sessions) with the Atalante device and 2 sessions per week (i.e., 12 one-hour sessions) of conventional therapy.
* For the Control group: 5 sessions per week of conventional therapy (i.e., 30 one-hour sessions).

The study will include 66 patients (33 in each arm) and takes place in two French centers, two German centers and one Spanish center.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* First clinically significant disability due to stroke
* Hemiparesis in acute-subacute phase (1 to 4 months since lesion) due to a stroke
* Functional Ambulation Category score (FAC) <2
* Patient with health insurance
* Informed and willing to sign an informed consent form approved by the Ethics Committee. For clarity, if a motor impairment prevents the subject from signing by himself, he/she can still be included if the signature can be done by an impartial witness.

Exclusion Criteria:

* Muscle overactivity in hip adductors, hamstrings, quadriceps and plantar flexors, which interferes with exoskeleton use, based on clinician investigator's opinion
* Recent fracture (< 3 months) or any therapy inducing secondary osteoporosis
* Excessive joint mechanical pain in the lower limbs based on clinician investigator's opinion
* Pressure sore grade I or more over contact zones with Atalante system, according to the International Pressure Ulcer Classification System NPUAP - EPUA
* Medical contra-indication to medium intensity physical strain
* Orthostatic hypotension (loss of > 20 mmHg systolic BP after 3 minutes in standing position)
* Uncontrolled seizures
* Morphological contra-indications to the use of Atalante (as per user's manual)
* Pregnant woman
* Adults who lack the capacity to provide informed consent, and all those persons deprived of their liberty in prisons or other places of detention
* Concurrent participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2023-06-12 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Walking recovery expressed by the proportion of patients reaching a Functional Ambulation Category (FAC) score of 4 or higher at the end of the intervention period, assessed without the exoskeleton. | End of the intervention period (week 6)
  The FAC is a 6-item ordinal scale that classifies the level of support needed to walk safely, irrespective of the use of a lower extremity orthosis or walking aid, ranging from 0 (unable to walk without the assistance of two people) to 5 (independent walking on uneven surfaces and on stairs).

SECONDARY OUTCOMES:
Walking recovery expressed by the proportion of patients reaching a FAC score of 4 or higher at six months post stroke, assessed without the exoskeleton. | 6 months post stroke
Time to reach FAC score of 4 or higher | Day 1 (± 3 days), week 2 (± 3 days) and week 4 (± 3 days) after the beginning of the intervention period, end of the intervention period (Week 6 ± 3 days), discharge from hospital and 6 months post stroke (± 6 days).
Change in walking speed measured with the 10 Meter Walk Test (10MWT) | Day 1 (± 3 days), end of the intervention period (Week 6 ± 3 days), discharge and 6 months post stroke (± 6 days)
  The 10MWT is used to assess gait speed in meters/second over a short distance. Two tests are successively administered, barefoot, at comfortable then at maximal walking speed without walking aids. If a patient is unable to ambulate at all, a score of 0 m/s is documented.
Changes in static and dynamic balance measured by the Berg Balance Scale (BBS) | Day 1 (± 3 days), end of the intervention period (Week 6 ± 3 days), discharge and 6 months post stroke (± 6 days)
  The BBS is a subjective, ordinal scale that assesses the ability to safely balance and avoid falls, during a series of functional tasks. It is thus also a measure of the amount of assistance needed to perform these tasks safely. In most items, the subject must maintain a given position for a specified time or complete moving tasks of varying difficulty. Subject receives a score from 0-4 at each of the 14 items on the ability to meet these balance dimensions.
Change in transfer time from wheelchair to toilet and back to wheelchair | Day 1 (± 3 days), end of the intervention period (Week 6 ± 3 days), discharge and 6 months post stroke (± 6 days)
  The purpose is to record the time needed by the patient to do the transfer wheelchair /toilet seat/ wheelchair. Reduction of this time could mean an improvement of independence in daily life for stroke patients for whom transferring to the toilet is a common difficulty.
Changes in maximal clinical muscle extensibility XV1 and maximal range of active motion XA against the resistance of the key lower limb muscles using the Five Step Assessment | Day 1 (± 3 days), end of the intervention period (Week 6 ± 3 days), discharge and 6 months post stroke (± 6 days)
  Measurements of XV1 and XA for soleus, gastrocnemius, gluteus maximus, hamstrings, vastus and rectus femoris muscles, using to the Five Step Assessment
  * XV1 is the angle of arrest at slow speed of stretch, corresponding to the passive range of motion against the resistance of the tested muscle.
  * XA is the maximal active range of motion against the resistance of the evaluated antagonist muscle.
Changes in anxiety and depression scores using the Hospital and Depression scale (HAD) | Day 1 (± 3 days), end of the intervention period (Week 6 ± 3 days), discharge and 6 months post stroke (± 6 days)
  The HAD is a two-dimension self-administered questionnaire developed to identify depression and anxiety among physically ill patients. Identifying these disorders and the context in which they develop is interesting as motivation of the patient seems to have an important impact on his progression. It consists of 14 items rated with a score from 0-4, divided into 7 items for anxiety and 7 items for depression based on the concept of anhedonia.
Changes in perceived quality of life assessed by the Short Form-36 (SF-36) | Day 1 (± 3 days) and 6 months post stroke (± 6 days)
  The SF-36 is a self-administered questionnaire that provides an evaluation of the generic Quality of Life. The version used is the RAND-36 Item Health Survey. There are 36 items (or questions) divided into eight domains:
  Physical component:
  1. Physical functioning
  2. Role limitations due to physical problems
  3. Bodily pain
  4. General health perceptions
     Mental component:
  5. Social functioning
  6. General mental health
  7. Role limitations due to emotional problems
  8. Vitality Each item is answered by the subject with a Likert scale.
Subject and Therapist satisfaction and willingness to continue training sessions | End of Week 1 (± 3 days), end of Week 3 (± 3 days) and end of the intervention period (Week 6 ± 3 days)
  The subject is asked to answer two questions regarding his satisfaction and willingness to continue training sessions. The therapist answers one question on his satisfaction. The score of each question is evaluated with a 5-level Likert scale.
Perceived workload by the therapists conducting sessions assessed with the NASA Task Load Index | End of Week 1 (± 3 days) and end of the intervention period (Week 6 ± 3 days)
  The NASA Task Load Index is a multidimensional, subjective scale that rates perceived workload in order to assess a task.There are six items, answered by the therapists after the therapy session:
  1. Mental demand
  2. Physical demand
  3. Temporal demand
  4. Effort
  5. Performance
  6. Frustration level The therapist gives his answers for the task "conducting a therapy session with the Atalante device" for patients of the Exo group, and for the task "conducting a conventional therapy session" for patients of the Control group.

CONTACTS AND LOCATIONS:
Locations (5):
- France (2):
  - Hôpitaux Universitaires Henri Mondor APHP, site Albert Chenevier, Créteil
  - Centre de Médecine Physique et de Réadaptation APAJH de Pionsat, Pionsat
- Germany (2):
  - Schön Klinik, Bad Aibling
  - Vivantes Klinikum Spandau, Berlin
- Institut Guttmann, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No